CLINICAL TRIAL: NCT06009939
Title: Microvascular Sex and Age-related Day-to-day Variability in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Vårdcentralen Åby (Other)
Collaborators: Department of Biomedical Engineering (IMT) (Unknown); Department of Health, Medicine and Caring Sciences (HMV) (Unknown); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Fredrik Iredahl, Associate Professor, Vårdcentralen Åby
Other Study IDs: 2023-01
Record Dates: First submitted 2023-08-09; First posted 2023-08-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy men aged 20-30 years old: Foot: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Arm: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Interventions: Other: Occlusion of the circulation in the arm and foot
- Healthy women aged 20-30 years old: Foot: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Arm: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Interventions: Other: Occlusion of the circulation in the arm and foot
- Healthy men aged 50-60 years old: Foot: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Arm: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Interventions: Other: Occlusion of the circulation in the arm and foot
- Healthy women aged 50-60 years old: Foot: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Arm: 10 minutes of baseline measurement, 5 minutes of occlusion and 5 minutes of Post-occlusive reactive hyperemia (PORH) measurement.
  Interventions: Other: Occlusion of the circulation in the arm and foot

INTERVENTIONS:
Other: Occlusion of the circulation in the arm and foot — A blood pressure cuff occludes the circulation in the upper arm as well as around the ankle.

SUMMARY:
The goal of this observational study is to learn more about the microcirculation in the skin by examining sex and age-related day-to-day variability in healthy subjects. The main questions the trial aims to answer are:

* What is the day-to-day variability of the optical measurement techniques in the microcirculation, and does age and gender affect this?
* Does the day-to-day variability differ in the foot compared to the arm?

Participants will rest whilst skin measurement by optical measurement techniques are performed. Baseline measurements and post-occlusive reactive hyperemia will be studied on the forearm and foot. This measurement procedure is repeated within one week, in order to study variability.

DETAILED DESCRIPTION:
The microcirculation consists of arterioles, capillaries and venules and is essential for nutrients and oxygen to be delivered to the tissue as well as waste products to be removed. The skin is often used as a model for studying microcirculation.

There are many different ways to study the microcirculation, most commonly are noninvasive optical techniques which measures the reflection of light used. Laser Doppler Flowmetry (LDF) has been the golden standard, but one limitation with the technique is that it measures the bloodflow in a small area (about 1 mm3). In this study the investigators will be using single-point measurement with a technique called EPOS and larger area measurements with a technique called PSI-X. EPOS, based on LDF and diffuse reflectance spectroscopy (DRS), analyze speed-resolved perfusion, variations in red blood cell tissue fraction, oxygen saturation and vessel diameter. PSI-X, based on multi-exposure laser speckle contrast imaging (MELSCI) and multispectral imaging (MSI), analyze conventional perfusion, speed-resolved perfusion and oxygen saturation.

Flowmotion is the rhythmical variations in measured skin blood flow that arise due to global and local regulation of the vessels and can be studied using frequency analysis of time-resolved blood flow signals. Since EPOS and PSI-X collect data of time-resolved blood flow, flowmotion analysis will also be conducted in the study.

To study day-to-day variability, data will be collected from each subject on two separate days within seven days, on the same location of the foot as well as the arm. Once the subject arrives to the lab, a questionnaire will be filled in regarding the subjects physical activity level, exercise habits and usage of medication and nicotine. The subject will also confirm to not have eaten two hours and not used nicotine or caffeine three hours prior to the experiment. Thereafter the subject's length and weight will be measured and BMI calculated. The subjects skin type will be determined using the Fitzpatrick scale. All of this is only done on the first day of measurement, on the second day the subject will skip right to the following part.

An acclimatization period of 15 minutes begins and the subject will remove socks and lay down. While the subject rests the equipment will be set up. A blood pressure cuff is placed around the upper arm as well as around the ankle. An EPOS-probe is placed on the dorsal side of the foot as well as the volar side of the forearm. A marker pen is used to mark the skin around the probes which enables the probe to be placed on the same location on the next measurement. Once five minutes has passed, the subject's blood pressure and pulse is noted. Thereafter the PSI-X camera is set up and angled to film the plantar side of the foot from a distance of about 25 cm. The subject is asked to lay as still as possible during the measurement. Once the acclimatization period has passed, the lights in the lab are turned off and the measurement will begin. Firstly baseline data will be collected as the subject rest for 10 minutes without provocation. Thereafter the blood pressure cuff on the ankle will inflate to 250 mmHg for five minutes whilst data is collected. Lastly data is collected for five minutes after the blood pressure cuff deflates. Thereafter the PSI-X camera is moved and angled to film the forearm from a 25 cm distance. The protocol described above is repeated for the arm. The subject will return within seven days to repeat the data collection protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20-30 years old and 50-60 years old

Exclusion Criteria:

* Regular use of medication (except for anti-conception medication)
* Hypertension
* Skin- or cardiovascular disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the investigators aim to study potential differences between men and women an equal number of men and women needs to be included in the study.
Study Population: 12 healthy men and 12 healthy women aged 20-30 years old. 12 healthy men and 12 healthy women aged 50-60 years old.
  In total 48 participants will be included.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Speed-resolved perfusion | Measured during 45 minutes and at one more occasion for 45 minutes within one week.
  [% RBC ×mm/s]
Red blood cell tissue fraction | Measured during 45 minutes and at one more occasion for 45 minutes within one week.
  [% RBC]
Oxygen saturation | Measured during 45 minutes and at one more occasion for 45 minutes within one week.
  [% oxygen]
Vessel diameter | Measured during 45 minutes and at one more occasion for 45 minutes within one week.
  [μm]

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Iredahl, Principal Investigator — Linköping University, Department of Health, Medicine and Caring Sciences
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Background] Hultman M, Larsson M, Stromberg T, Henricson J, Iredahl F, Fredriksson I. Flowmotion imaging analysis of spatiotemporal variations in skin microcirculatory perfusion. Microvasc Res. 2023 Mar;146:104456. doi: 10.1016/j.mvr.2022.104456. Epub 2022 Nov 18. No abstract available. PMID 36403668
- [Background] Fredriksson I, Larsson M, Stromberg T, Iredahl F. Vasomotion analysis of speed resolved perfusion, oxygen saturation, red blood cell tissue fraction, and vessel diameter: Novel microvascular perspectives. Skin Res Technol. 2022 Jan;28(1):142-152. doi: 10.1111/srt.13106. Epub 2021 Nov 10. PMID 34758168
- [Background] Hultman M, Larsson M, Stromberg T, Fredriksson I. Real-time video-rate perfusion imaging using multi-exposure laser speckle contrast imaging and machine learning. J Biomed Opt. 2020 Nov;25(11):116007. doi: 10.1117/1.JBO.25.11.116007. PMID 33191685
- [Background] Hultman M, Larsson M, Stromberg T, Fredriksson I. Speed-resolved perfusion imaging using multi-exposure laser speckle contrast imaging and machine learning. J Biomed Opt. 2023 Mar;28(3):036007. doi: 10.1117/1.JBO.28.3.036007. Epub 2023 Mar 20. PMID 36950019

DOCUMENTS (2):
  • Study Protocol (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT06009939/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT06009939/SAP_001.pdf